CLINICAL TRIAL: NCT00767546
Title: Botulinum Toxin for Treatment of Seborrhic Dermatitis in Parkinsonian Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr Joseph Zoldan, Neurology department, Rabin medical center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004988
Record Dates: First submitted 2008-10-05; First posted 2008-10-07 (Estimated); Last update posted 2008-10-07 (Estimated); Status verified 2008-10

CONDITIONS: Parkinson Disease; Parkinsonism; Seborrheic Dermatitis
Keywords: seborrhic dermatitis; parkinson's disease; Parkinson disease parkinsonism and seborrhic dermatitis
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Dermatitis, Seborrheic | interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinum toxin — 60- 100 units Local injection to the rash area

SUMMARY:
There's high incidence of seborrhic dermatitis among patients suffering from Parkinson's disease. Seborrhic dermatitis is caused by increased exertion of sebaceous glands. Previous studies have shown an increase of sebum excretion rate in parkinsonian pateints. Other studies demonstrated improvement in seborrhic dermatitis after anticholinergic treatment. From these studies we concluded that there might be hyperactivity of the parasympathetic system among PD patients, that cause increased exertion of sebum, therefore local injection of botulinium toxin, which inhibitis acetyl choline realese, might improve the rash of seborrhic dermatitis.

40 patients suffering from Parkinson disease or other parkinsonian disorders will participate in this study.

Before treating the patients with botulinium toxin, we will measure the sebum exertion with the sebumeter device and make clinical evaluation of the rash. We will also take a picture of the rash.

Then Botulinium toxin (60- 100 units) will be locally injected to the rash area.

Two weeks after the injection the patients will be called and evaluated clinicly and by the sebumeter. Then they will be checked again after 3 weeks, after a month and after two, three and four month's.

DETAILED DESCRIPTION:
Exclusion criteria:

* Dementia
* Renal or liver failure
* Pregnancy or breast feeding
* History of allergy to botolinium toxin
* Motor neuron disease or any other disease that insult the neuromuscular junction
* Treatment with Amynoglycoside antibiotic. This study will include only patients that can give informed concent.

SEBUMETER SM 810- this is the device we will use to measure sebum exertion before and after injecting botulinium toxin. The measurement is based on grease-spot photometry. A special tape becomes transparent in contact with the sebum on the skin surface. For the determination of the sebum, the measuring head of the cassette is inserted into the aperture of the device, where the transparency is measured by a light source sending light through the tape which is reflected by a little mirror behind the tape. A photocell measures the transparency. The light transmission represents the sebum content on the surface of the measuring area. A microprocessor calculates the result, which is shown on the display in µg sebum/cm² of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease patients that have seborrhic dermatits

Exclusion Criteria:

* Dementia
* Renal or liver failure
* Pregnancy or breast feeding
* History of allergy to botolinum toxin
* Motor neuron disease or any other disease that insult the neuromuscular junction
* Treatment with Aminoglycoside antibiotic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Clinical assesment of the rash Photometric test of sebum exertion | 4 month